CLINICAL TRIAL: NCT06295406
Title: Reading Ability in Childhood Obesity
Acronym: Lettura_evOB
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 21C310
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Obesity, Childhood; Obesity, Adolescent
Keywords: Reading abilities; Cognitive functioning; Neuropsychological assessment; Motor abilities
MeSH Terms: conditions — Pediatric Obesity | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Participants with age range between 11 and 16 years, with overweight (BMI>85° ) or obesity (BMI>95°)
  Interventions: Other: Neuropsychological assessment

INTERVENTIONS:
Other: Neuropsychological assessment — Neuropsychological tests assessing reading abilities, skills of motor coordination, postural stability, manual dexterity, including graphomotor skills, and estimation of time will be performed

SUMMARY:
There is some evidence about the negative impact of overweight and obesity on reading ability, with negative consequences on quality of life and school success.

In this neuropsychological research, the relationship between the characteristics of reading abilities in individuals with obesity (age range between 11 and 16 years) and the skills of motor coordination, postural stability, manual dexterity, including graphomotor skills, and estimation of time is investigated according to the cerebellar deficit theory.

ELIGIBILITY:
Inclusion criteria

• diagnosis of overweight or obesity

Exclusion criteria:

• concurrent neurological, neurodevelopmental (e.g., autism), motor, somatosensory and/or psychiatric disorders.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants with obesity will be recruited at the beginning of a rehabilitative treatment at the Istituto Auxologico Italiano, IRCCS, San Giuseppe Hospital (Italy).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Raw score at the neuropsychological assessment | baseline
  For each neuropsychological test, the raw score reported by the participants will be computed according to the validation norms. There are different levels of minumun and maximum scores for each neuropsychological tests.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Auxologico Italiano - Ospedale San Giuseppe, Piancavallo, VCO, Italy